CLINICAL TRIAL: NCT01662973
Title: Phase 1/2 Study of UC-MSC Treatment for Evaluation the Efficacy and Safety in Patients With Primary Biliary Cirrhosis
Brief Title: Umbilical Cord Mesenchymal Stem Cells for Patients With Primary Biliary Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Director of both the Research Center for Biological Therapy and the Beijing Institute of Translational Hepatology, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302-005
Record Dates: First submitted 2012-08-05; First posted 2012-08-13 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis; Mesenchymal Stem Cells; Serum alkaline phosphatase; Serum Bilirubin
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional plus UC-MSC treatment (Experimental): Participants will receive conventional treatment plus a dose of UC-MSC from day 0 through the week 12 study visit.
  Participants will then be followed until the week 48 study visit.
  Interventions: Other: conventional plus UC-MSC treatment
- Conventional plus placebo treatment (Placebo Comparator): Participants will receive conventional plus placebo treatment from day 0 through the week 12 study visit. Participants will then be followed until the week 48 study visit.
  Interventions: Other: Conventional plus placebo treatment

INTERVENTIONS:
Other: conventional plus UC-MSC treatment — Received conventional treatment and taken i.v., once per 4 week, at a dose of 1*10E6 UC-MSC/kg body weight for 12 weeks.
  Arms: Conventional plus UC-MSC treatment
Other: Conventional plus placebo treatment — Received conventional treatment and taken i.v., once per 4 week, at 50 ml saline for 12 weeks
  Arms: Conventional plus placebo treatment

SUMMARY:
Primary biliary cirrhosis (PBC) is a slowly progressive disease that causes substantial loss of intrahepatic bile ducts, ultimately resulting in cholestasis, advanced fibrosis, cirrhosis, liver failure and even hepatocellular carcinoma. Histologically, the disease is characterized by chronic portal inflammation with infiltration, destruction and loss of the epithelial cells in the small-sized and medium-sized bile ducts. Currently, Ursodeoxycholic acid (UDCA) in a dose of 13-15mg/kg/day is recommended as therapeutic drugs for PBC by AASLD and is approved for this indication by the U.S. Food and Drug Administration (FDA). Treatment with UDCA may delay disease progression and prolong survival free of liver transplantation. However, one out of three patients does not adequately respond to UDCA therapy and many need additional medical therapy or liver transplantation, or both. UC-MSC has been application for the treatment of several severe autoimmune diseases, such as immune thrombocytopenia, systemic lupus erythematosus, and therapy-resistant rheumatoid arthritis. In this study, the safety and efficacy of UC-MSC transplantation for PBC patients will be evaluated.

DETAILED DESCRIPTION:
Primary biliary cirrhosis (PBC) is a slowly progressive cholestatic disease associated with the development of cirrhosis and liver failure that may justify liver transplantation. Ursodeoxycholic acid (UDCA) is currently the only drug approved specifically for the treatment of PBC. However, one out of three patients does not adequately respond to UDCA therapy and many need additional medical therapy or liver transplantation, or both.

The potential for stem cells to differentiate into biliary epithelial cells was recently confirmed. In particular, bone marrow-derived mesenchymal stem cell (BM-MSC) transplantation has been applicated in the clinic for treat several human disease such as GVHD, cardiac injury and brain injury, and displayed good tolerance and efficiency. Recently, umbilical cord-derived MSCs (UC-MSC) has also been used to treat severe autoimmune diseases, such as therapy-resistant rheumatoid arthritis and multiple sclerosis.

The purpose of this study is to learn whether and how UC-MSC can improve the disease condition in patients with primary biliary cirrhosis. This study will also look at how well UC-MSC is tolerated and its safety in PBC patients

Participants in the study will be randomly assigned to one of two treatment arms:

Arm A: Participants will receive 12 weeks of UC-MSC treatment plus UDCA. Arm B: Participants will receive 12 weeks of placebo plus UDCA. UC-MSC will be prepared according to standard procedures and is collected in plastic bags containing anticoagulant. UC-MSCs are given via i.v. under sonography monitoring. After cell therapy, patients are followed up at week 4,8,12,24,36 and 48. The evaluation of some clinical parameters such as the level of serum alkaline phosphatase (ALP), alanine aminotransferase(ALT) aspartate aminotransferase (AST) and total bilirubin (TB), prothrombin time(PT), albumin(ALB), prealbumin(PA), are detected at these time points. Mayo risk score, portal hypertension, Liver histology, MELD score and clinical symptoms were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Primary Biliary Cirrhosis (according to the criteria defined by AASLD practice guidelines , Hepatology, 2009;50:291-308 )
3. Negative pregnancy test (female patients in fertile age)

Exclusion Criteria:

1. Hepatocellular carcinoma or other Malignancies
2. Pregnant or lactating women
3. Viral Hepatitis ( HAB, HBV, HCV, et al )
4. Vital organs failure (Cardiac, Renal or Respiratory, et al)
5. Sepsis
6. Active thrombosis in the portal or hepatic veins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Serum alkaline phosphatase (ALP) | 0, 4, 8,12, 24, 36,48 weeks after treatment

SECONDARY OUTCOMES:
Histological changes in liver biopsies | baseline and 48 weeks
Serum Bilirubin | At base line and at week 4,8,12,24,36 and 48
Serum AST | At base line and at week 4,8,12,24,36 and 48
Mayo risk score | At base line and at week 4,8,12,24,36 and 48
Number of patients with Portal Hypertension after 12 weeks treatment | At base line and at week 12,24,36 and 48
MELD score | At base line and at week 4,8,12,24,36 and 48
Number of participants with improvement of clinical symptoms | At base line and at week 4,8,12,24,36 and 48
  clinical symptoms including fatigue (Fatigue Impact Score, FIS) and pruritus ( Visual Analog Scale ,VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, professor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Poupon RE, Lindor KD, Cauch-Dudek K, Dickson ER, Poupon R, Heathcote EJ. Combined analysis of randomized controlled trials of ursodeoxycholic acid in primary biliary cirrhosis. Gastroenterology. 1997 Sep;113(3):884-90. doi: 10.1016/s0016-5085(97)70183-5. PMID 9287980
- [Background] Kuiper EM, Hansen BE, de Vries RA, den Ouden-Muller JW, van Ditzhuijsen TJ, Haagsma EB, Houben MH, Witteman BJ, van Erpecum KJ, van Buuren HR; Dutch PBC Study Group. Improved prognosis of patients with primary biliary cirrhosis that have a biochemical response to ursodeoxycholic acid. Gastroenterology. 2009 Apr;136(4):1281-7. doi: 10.1053/j.gastro.2009.01.003. Epub 2009 Jan 14. PMID 19208346
- [Background] Poupon R. Primary biliary cirrhosis: a 2010 update. J Hepatol. 2010 May;52(5):745-58. doi: 10.1016/j.jhep.2009.11.027. Epub 2010 Feb 18. PMID 20347176
- [Background] Silveira MG, Brunt EM, Heathcote J, Gores GJ, Lindor KD, Mayo MJ. American Association for the Study of Liver Diseases endpoints conference: design and endpoints for clinical trials in primary biliary cirrhosis. Hepatology. 2010 Jul;52(1):349-59. doi: 10.1002/hep.23637. No abstract available. PMID 20578151